CLINICAL TRIAL: NCT05230004
Title: Innovative Prosthetic Systems for Pediatric Limb Loss to Accommodate Growth
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Children's Hospital of Philadelphia (Other)
Responsible Party: Principal Investigator, Timothy Dillingham, The William J. Erdman II, Professor and Chair, University of Pennsylvania
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 849980
Record Dates: First submitted 2022-01-13; First posted 2022-02-08 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: Limb Deficiencies; Pediatric ALL
Keywords: prosthesis; limb deficiency; limb loss; pediatric
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Phase II (Experimental): Phase II involves a two month home trial to determine the comfort and utility of an adjustable prosthetic system for children. Children will be fit at several different locations by their prosthetist with the adjustable socket. They will complete several questionnaires on their current device, as well as have internal socket pressures and a gait analysis completed. They will return one month later to complete the same outcome measures on their conventional device. They will also be given activity monitors to track their activity through the duration of the project.
  Interventions: Device: iFIT prosthesis
- Phase I (Experimental): Phase I involves developing a final design for an adjustable, immediate fit prosthesis. We will recruit 5-10 participants age 3-12 to complete in-lab testing and evaluation of several designs. This testing will lead to the final product design to be tested in Phase II.
  Interventions: Device: iFIT prosthesis

INTERVENTIONS:
Device: iFIT prosthesis — An adjustable modular prosthesis that can be fit in a single session. Fully adjustable by wearer.

SUMMARY:
An immediate fit adjustable prosthetic system is being investigated for children. The age range being recruited is from 3 years up to 18 years old. Phase I of this study will involve developing a final prototype by conducting in-lab testing on children with limb loss. Phase II will involve a two month home trial to further evaluate the comfort and usability of the socket. Outcome measures include a PEQ-based questionnaire, socket pressure measures and gait analysis.

DETAILED DESCRIPTION:
Design Phase I is a testing session to obtain feedback on initial prototype designs for the immediate fit prostheses. This research will focus on PI observations and participant feedback through survey and comments during the in-person testing. There may be multiple appointments for participants during this time the device design is refined. In-lab testing only will occur. This information will influence the overall design of the final prosthesis.

PHASE I: For Phase I children with lower limb limb loss (below the knee or above the knee) age 3-12 are being recruited. Subjects should be able to ambulate with or without assistive devices. They will supply measurements and limb images prior to the appointment.

During the initial appointment, each participant will be consented and completed roughly 2-3 hours of device testing. The participant will be fit with an adjustable prosthetic by the PI. After ambulating in the lab, they will give feedback on the comfort, stability and ease of use of the prosthesis. Participants may be asked to return several times for future testing sessions once changes or alterations are made to the prosthesis design to see if these have been effective. The child and their parent will fill out a PEQ based questionnaire on their conventional prosthesis and the investigational device after fitting.

Phase II: We will be recruiting children ages 3-18 with lower limb loss to be with an adjustable prosthesis and wear it for a 2 month home trial. Children may be recruited at other locations such as the Children's Hospital of Philadelphia and Ai./duPont Nemours in Delaware. The child and their parent will fill out questionnaires on their current prosthesis as well as have pressure data and a gait analysis completed. Once they have worn the prosthesis for 2 months they will return and complete these same outcome measures.

Gait biomechanical analysis: This analysis will be conducted by having several reflective markers placed on the participant's lower body. The subject will then walk a minimum of 6 times along a 10meter walkway while being recorded by the motion analysis system. This will be conducted in both the adjustable and conventional prosthesis.

Internal pressure measurements of the socket using Fujifilm pressure paper will also be obtained. Five spots will be assessed by placing the paper on the participant's liner and then they will put on their socket and walk for 1 minute. This will be completed on both the test and conventional socket.

ELIGIBILITY:
Inclusion Criteria:

* Four months post-amputation
* Subjects who have lost a limb due to any cause: trauma, congenital limb loss, dysvascular causes (peripheral vascular disease and diabetes), or malignancy will all be eligible for inclusion.
* Intact, protective sensation in their residual limbs.

Exclusion Criteria:

* open skin lesions
* excessive pain in the residual limb (phantom pain, residual limb pain, or neuroma)
* neurological disorders (e.g., stroke, severe polyneuropathy) causing weakness in the contralateral leg or marked gait impairment
* inability to follow instructions for trial

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 28 (Actual)
Dates: Start 2022-08-18 (Actual); Primary Completion 2025-03-07 (Actual); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Modified Prosthetic Evaluation Questionnaire | 2 months
  Evaluation questionnaire for prosthesis. Questions selected from PEQ are rated from 1-poor, to 5 excellent. 70 points total
Internal Socket Pressures | 2 months
  Fujifilm pressure paper will be taped to the inside of the conventional socket and test socket to determine internal pressure values. Participants will walk at a self selected walking speed for 30 seconds.
Socket Comfort Score | 2 months
  Rating of socket comfort from 0 very uncomfortable to 10 very comfortable
Gait Speed | 2 months
  Participants will walk at a self-selected walking speed while being recorded by 3d motional analysis cameras. They will walk across a 10 meter runway six times in their conventional socket and six times in the test socket to determine average walking speed.
PedsQL | 2 months
  quality of life survey for children
CAPP-PSI | 2 months
  brief, parent-administered inventory for the assessment of prosthesis satisfaction in children with limb deficiency.

CONTACTS AND LOCATIONS:
Overall Officials: Timothy R Dillingham, MS,MD, Principal Investigator — University of Pennsylvania
Locations (1):
- Penn Medicine Rittenhouse, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McCloskey C, Kenia J, Shofer F, Marschalek J, Dillingham T. Improved Self-Reported Comfort, Stability, and Limb Temperature Regulation with an Immediate Fit, Adjustable Transtibial Prosthesis. Arch Rehabil Res Clin Transl. 2020 Dec;2(4):100090. doi: 10.1016/j.arrct.2020.100090. Epub 2020 Nov 2. PMID 33381750
- [Background] Kenia J, Wolf B, Marschalek J, Dillingham T. An Immediate Fit, Adjustable, Modular Prosthetic System for Addressing World-Wide Limb Loss Disability. Arch Rehabil Res Clin Transl. 2021 Mar 15;3(2):100120. doi: 10.1016/j.arrct.2021.100120. eCollection 2021 Jun. PMID 34179756
- See also: This is the website for the adult adjustable prosthetic system — http://www.ifitprosthetics.com